CLINICAL TRIAL: NCT01276184
Title: A Randomized, Controlled Trial to Compare the Effectiveness of SMS Text Message Reminders Compared to Usual Care to Increase Adherence to the Gardasil Vaccine Dosing Schedule (GCC 1063GCC).
Brief Title: Effectiveness of SMS (Short Message Service) Text Messaging in Increasing Adherence to Gardasil
Acronym: CHAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient sample for study completion.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, J. Kathleen Tracy, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HP-00047046; GCC 1063GCC (Other: GCC accession number); Merck-37944 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: HPV Vaccines
Keywords: HPV Vaccine; HPV vaccination; SMS; Text Message; Gardasil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants follow the usual practices for scheduling their follow up visit(s) for vaccination at the clinic. Participants will receive the standard reminder from the clinic for their scheduled appointment(s) (phone call, letter, etc, as appropriate).
- SMS Text Message (Experimental): Participants in both the Usual Care group and the SMS Text Message group will receive the standard reminder from the clinic for their scheduled appointment(s) (phone call, letter, etc, as appropriate). Women in the SMS Text Message group that reschedule a vaccination visit will receive text message reminders one per day for each of the seven days prior to the rescheduled visit.
  Interventions: Behavioral: SMS Text Message

INTERVENTIONS:
Behavioral: SMS Text Message — Women in the SMS Text Message group that reschedule a vaccination visit will receive text message reminders one per day for each of the seven days prior to the rescheduled visit (or as many days as possible depending on when the rescheduled visit will take place - for example, if they call in and reschedule the visit to take place in 4 days, they will receive text messages for the 3 days prior to the rescheduled visit). Participants in both the Usual Care group and the SMS Text Message group will receive the standard reminder from the clinic for their re-scheduled appointment(s).
  Other Names: Usual care; Text message
  Arms: SMS Text Message

SUMMARY:
Human papillomavirus (HPV) is the most common sexually transmitted disease among adolescent females in the United States. Our primary objective is to determine if Short Message Service (SMS) text message reminders increase adherence to the recommended 3 dose schedule for Gardasil compared to usual care in an outpatient clinic setting. Secondary objectives of this study are: 1) to demonstrate the feasibility of using SMS text message reminders to increase adherence with Gardasil vaccination; and 2) to assess satisfaction and acceptability of text message reminders compared to telephone reminders among women who receive the text message arm of the intervention. The investigators hypothesize that receiving SMS text message reminders will increase adherence to the recommended 3 dose schedule for Gardasil compared to usual care.

DETAILED DESCRIPTION:
Technological innovations such as Short Message Service (SMS) text messages reminders are one strategy that may be used to increase adherence to the Gardasil dosing schedule. Although the literature in this area is in its infancy, several studies have demonstrated that SMS text reminders are an effective strategy for reducing nonattendance with medical appointments. Further, SMS text message reminders have been shown to be popular with patients and more cost-effective than paper or telephone-based reminder strategies. The investigators believe SMS text message reminders can be used as a feasible and cost-effective strategy to increase adherence to the Gardasil vaccine schedule, thus reducing risk of cervical cancer.

Women who are enrolled will be randomly assigned to one of 2 study groups (Usual Care v. SMS Text Message group). For women in the SMS Text Message group, text message reminders will be sent once per day for each of the seven days prior to the scheduled date for each of their follow up vaccinations. Participants follow the usual practices for scheduling their follow up visit(s) for vaccination at the clinic. Participants in both the Usual Care group and the SMS Text Message group will receive the standard reminder from the clinic for their scheduled appointment(s) (phone call, letter, etc, as appropriate). At enrollment, the participant will answer questions regarding social and demographic history, cell phone use patterns, attitudes and acceptance of HPV vaccine, gynecologic and sexual history.

All participants will be sent a packet of self-report measures to complete regarding attitudes toward HPV vaccination at the completion of the study. Participants in the SMS Text Message group will also receive rating scales to assess acceptability of text message reminders and preference for text message reminders over telephone reminders.

ELIGIBILITY:
Inclusion Criteria:

* Have a mobile phone with text message capability
* Patient of University of Maryland Medical Center outpatient gynecology clinics
* Able to speak and read English
* Capable of understanding, consenting, and complying with the entire study protocol

Exclusion Criteria:

* Pregnant
* Previously completed the Gardasil vaccine

Ages: 12 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Tracy, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - Redwood Clinic, Baltimore, Maryland
  - Western-Penn Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 participants recruited.
Groups:
- SMS Text Message: Participants in both Usual Care group and the SMS Text Message group will receive the standard reminder from the clinic for their scheduled appointment(s) (phone call, letter, etc, as appropriate). Women in the SMS Text Message group that reschedule a vaccination visit will receive text message reminders one per day for each of the seven days prior to the rescheduled visit.
  SMS Text Message: Women in the SMS Text Message group that reschedule a vaccination visit will receive text message reminders one per day for each of the seven days prior to the rescheduled visit (or as many days as possible depending on when the rescheduled visit will take place - for example, if they call in and reschedule the visit to take place in 4 days, they will receive text messages for the 3 days prior to the rescheduled visit). Participants in both the Usual Care group and the SMS Text Message group will receive the standard reminder from the clinic for their re-scheduled appointment(s) (phone call,
Period: Overall Study
Arm/Group | Usual Care | SMS Text Message
Started | 13 | 9
Completed | 13 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SMS Text Message: Participants in both Usual Care group and the Text Message group will receive the standard reminder from the clinic for their scheduled appointment(s). Women in the SMS Text Message group that reschedule a vaccination visit will receive text message reminders one per day for each of the seven days prior to the rescheduled visit.
  SMS Text Message: Women in the SMS Text Message group that reschedule a vaccination visit will receive text message reminders one per day for each of the seven days prior to the rescheduled visit (or as many days as possible depending on when the rescheduled visit will take place - for example, if they call in and reschedule the visit to take place in 4 days, they will receive text messages for the 3 days prior to the rescheduled visit). Participants in both the Usual Care group and the SMS Text Message group will receive the standard reminder from the clinic for their re-scheduled appointment(s) (phone call, letter, etc, as appropriate).
- Total: Total of all reporting groups
Arm/Group | Usual Care | SMS Text Message | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 11 | 7 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 19 [12 to 26] | 17 [12 to 26] | 18 [12 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Adhered to Vaccine Schedule
Description: Our primary objective is to determine if Short Message Service (SMS) text message reminders increase number of participants that adhered to the recommended 3 dose schedule for Gardasil compared to usual care in an outpatient clinic setting.
Time Frame: at the end of the study (30 days after the third vaccination or 360 days after the first vaccination, whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | SMS Text Message
Number analyzed (Participants) | 13 | 9
Participants | 10 | 8

ADVERSE EVENTS:
Groups:
- SMS Text Message: Participants in both Usual Care group and the SMS Text Message group will receive the standard reminder from the clinic for their scheduled appointment(s) (phone call, letter, etc, as appropriate). Women in the SMS Text Message group that reschedule a vaccination visit will receive text message reminders one per day for each of the seven days prior to the rescheduled visit.
  SMS Text Message: Women in the SMS Text Message group that reschedule a vaccination visit will receive text message reminders one per day for each of the seven days prior to the rescheduled visit (or as many days as possible depending on when the rescheduled visit will take place - for example, if they call in and reschedule the visit to take place in 4 days, they will receive text messages for the 3 days prior to the rescheduled visit). Participants in both the Usual Care group and the SMS Text Message group will receive the standard reminder from the clinic for their re-scheduled appointment(s).
Arm/Group | Usual Care | SMS Text Message
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No